CLINICAL TRIAL: NCT05883982
Title: Analysis of the Results of Treatment With Intra-articular I-PRF Injections in Patients With Temporomandibular Joint Dysfunction.
Brief Title: Intra-articular I-PRF Injections in Patients With Temporomandibular Joint Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital of the Ministry of Interior, Kielce, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/2022/1
Record Dates: First submitted 2023-05-22; First posted 2023-06-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: We do not choose to create a placebo group or treatment groups other than intra-articular injections. In qualified patients, the administration of the substance into the temporomandibular joint cavity will be the treatment of choice or the generally accepted continuation of therapy in which the first-line treatment (pharmacotherapy, physiotherapy, splint therapy) turned out to be ineffective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- I-PRF (Experimental): Patients receiving I-PRF injections into temporomandibular joints.
  Interventions: Procedure: I-PRF injection

INTERVENTIONS:
Procedure: I-PRF injection — Intra-articular I-PRF injection to temporomandibular joint cavity

SUMMARY:
The aim of the study will be to analyze the results of injection treatment in patients diagnosed with temporomandibular joint dysfunction manifested by pain and/or limited jaw mobility. The treatment will consist in the administration of autologous blood products into the cavities of the temporomandibular joints.

DETAILED DESCRIPTION:
The aim of the study is to analyze the results of injection treatment in patients diagnosed with temporomandibular joint dysfunction manifested by pain and/or limited jaw mobility. The analyzed treatment will consist in the administration of autologous blood products into the cavities of the temporomandibular joints. We intend to conduct a prospective study without a control group. Patients suffering from pain in the temporomandibular joints and/or limited jaw mobility, in whom injection treatment is the treatment of choice, and patients in whom first-line therapies (pharmacotherapy, physiotherapy, splint therapy) did not bring the desired results, and intra-articular injections are a generally accepted continuation of the therapeutic protocol. Qualified patients will be treated with autologous blood products (injectable platelet-rich fibrin). Data from specialist literature support the safety and effectiveness of administering the above-mentioned substance to the cavities of the temporomandibular joints. The use of blood products in the form of intra-articular injections is medically justified both in the case of pain in the temporomandibular joints and/or in clinical conditions with limited jaw mobility. Currently available scientific publications on the comparison of the effectiveness of therapy with the use of various autologous substances are not numerous and do not give a clear answer to the question of what therapeutic protocol (type of substance, dose, number of administrations, joint compartment) is the most effective in the given observation period. This study aims to clarify some of these issues in regard to the above-mentioned blood product, and thus to obtain valuable clinical data that may help clinicians in choosing the appropriate use of intra-articular injections in patients with temporomandibular joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* age over 18;
* informed consent to participate in the study;
* the possibility of discontinuing the current treatment of the temporomandibular joints;
* generally accepted indications for injection therapy.

Exclusion Criteria:

* bleeding diathesis;
* mental illness;
* temporomandibular joint prosthesis;
* temporomandibular joint ankylosis;
* skin disease of the preauricular area of the affected side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Articular pain | 0 - 6 months
  Temporomandibular joint pain intensity on Visual Analogue Scale (form "0" - no pain to "10" - worst pain)
Mandibular mobility | 0 - 6 months
  Range of mandibular abduction (between incisal edges, in mm)

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Sikora, dr hab., Study Chair — Hospital of the Ministry of Interior, Wojska Polskiego 51, 25-375 Kielce, Poland
Locations (1):
- Department of Maxillofacial Surgery, Kielce, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sielski M, Checinska K, Turosz N, Checinski M, Sikora M. Single intra-articular administration of injectable platelet-rich fibrin (I-PRF) in alleviating temporomandibular joint pain: A pilot clinical trial. Dent Med Probl. 2025 Jan-Feb;62(1):187-192. doi: 10.17219/dmp/188273. PMID 40043084